CLINICAL TRIAL: NCT03520192
Title: Critically Ill Children and Young People: do National Differences in
Brief Title: Differences in Access to Emergency Paediatric Intensive Care and Care During Transport
Acronym: DEPICT
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 15HC47
Record Dates: First submitted 2017-11-09; First posted 2018-05-09 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Access and Transport to Paediatric Intensive Care
Keywords: Paediatric; Critical care; Transport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are fewer than 30 paediatric intensive care units (PICUs) in the United Kingdom (UK). This means that a critically ill child taken to their nearest hospital will need to be transferred to a PICU. Such transports are usually done by PICU retrieval teams (PICRTs), mobile teams who take specialist expertise to the child and safely transport them to a PICU.

There are national variations in how PICRTs are organised and deliver clinical care. There has been little research into these differences and how they might influence outcomes and experiences for sick children and families. The investigators do not know if national variation in how PICRT services are organised and delivered matters, or whether current standards help achieve the best outcomes for patients. This clinical study aims to understand how existing differences in access to paediatric intensive care and care provided by PICRTs affect clinical outcomes and experiences for transported critically ill children and families. The investigators will analyse routine national audit data to examine various aspects such as how long it takes a PICRT to reach the patient, how long it takes the child to reach the PICU, the seniority of clinicians performing the transport, medical procedures performed by the PICRT and any critical incidents during transport, and investigate whether any of these factors influence how likely a child is to survive. The investigators will also collect and analyse information about the experiences of sick children by interviewing the families involved, and staff experiences of PICU retrieval by interviewing clinicians. Alongside this work, the investigators will look at the costs of different ways of delivering PICRT services for sick children, and use mathematical techniques to study if and how alternate models of service delivery can improve clinical outcomes in a cost effective manner. The research team in this trial includes PICU and transport clinicians, parents, academic experts and an National Health Service (NHS) commissioner.

Independent committees consisting of clinicians and parents will be formed to oversee the study. The work from this study will directly inform the development of evidence-based national standards for PICU transport and help improve the patient experience for critically ill children and their families.

ELIGIBILITY:
Inclusion Criteria:

* Children and young people (age <16 years) transported by a PIC retrieval team for emergency admission to a paediatric intensive care unit in England and Wales.

Exclusion Criteria:

* None

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and young people (age <16 years) transported by a PIC retrieval team for emergency admission to a paediatric intensive care unit in England and Wales.
Sampling Method: Non-Probability Sample
Enrollment: 2838 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Number

SECONDARY OUTCOMES:
Mortality | up to 90 days
  Number
Mortality | 90 days
  Number
Mortality | One year
  Number
Length of stay | up to 90 days
  Number (days)
Days on invasive ventilation | up to 90 days
  Number (days)
Vasoactive agent therapy | up to 90 days
  Number (days)
Renal replacement therapy | up to 90 days
  Number (days)
Extra-corporeal life support | up to 90 days
  Number (days)
Length of hospital stay | up to 90 days
  Number (days)
Number of hospital admissions | One year
  Number
Days in hospital | One year
  Number (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramnarayan P, Evans R, Draper ES, Seaton SE, Wray J, Morris S, Pagel C; DEPICT Study Investigators. Differences in access to Emergency Paediatric Intensive Care and care during Transport (DEPICT): study protocol for a mixed methods study. BMJ Open. 2019 Jul 16;9(7):e028000. doi: 10.1136/bmjopen-2018-028000. PMID 31315865
- [Result] Seaton SE, Ramnarayan P, Pagel C, Davies P, Draper ES; DEPICT Study Team. Impact on 30-day survival of time taken by a critical care transport team to reach the bedside of critically ill children. Intensive Care Med. 2020 Oct;46(10):1953-1955. doi: 10.1007/s00134-020-06149-5. Epub 2020 Jun 22. No abstract available. PMID 32572530
- [Result] Seaton SE, Ramnarayan P, Davies P, Hudson E, Morris S, Pagel C, Rajah F, Wray J, Draper ES; DEPICT Study Team. Does time taken by paediatric critical care transport teams to reach the bedside of critically ill children affect survival? A retrospective cohort study from England and Wales. BMC Pediatr. 2020 Jun 19;20(1):301. doi: 10.1186/s12887-020-02195-6. PMID 32560633
- [Result] Seaton SE, Draper ES, Pagel C, Rajah F, Wray J, Ramnarayan P; DEPICT Study Team. The effect of care provided by paediatric critical care transport teams on mortality of children transported to paediatric intensive care units in England and Wales: a retrospective cohort study. BMC Pediatr. 2021 May 3;21(1):217. doi: 10.1186/s12887-021-02689-x. PMID 33941116
- [Result] Evans REC, Barber V, Seaton S, Ramnarayan P, Davies P, Wray J; DEPICT Study Group. Is Parental Presence in the Ambulance Associated With Parental Satisfaction During Emergency Pediatric Intensive Care Retrieval? A Cross-Sectional Questionnaire Study. Pediatr Crit Care Med. 2022 Sep 1;23(9):708-716. doi: 10.1097/PCC.0000000000002995. Epub 2022 May 27. PMID 35969657
- [Result] Evans REC, Barber V, Seaton S, Draper ES, Rajah F, Pagel C, Polke E, Ramnarayan P, Wray J; DEPICT Study Investigators. Development of a parent experience measure for paediatric critical care transport teams. Nurs Crit Care. 2022 May;27(3):367-374. doi: 10.1111/nicc.12648. Epub 2021 May 24. PMID 34028143
- [Derived] Alexander EC, Mallick A, Seaton SE, Evans R, Barber V, Wray J, Ramnarayan P; Differences in Access to Emergency pediatric Intensive Care and care during Transport (DEPICT) study group. Child and Parent Outcomes in the 2018-2019 DEPICT (Differences in Access to Emergency Pediatric Intensive Care and Care During Transport) Study: 12-Month Follow-Up Data. Pediatr Crit Care Med. 2025 Dec 19. doi: 10.1097/PCC.0000000000003877. Online ahead of print. PMID 41416858